CLINICAL TRIAL: NCT01307332
Title: Advanced Magnetic Resonance Imaging Measures of Repair in Alemtuzumab Treated Patients
Brief Title: Advanced MRI Measures of Repair in Alemtuzumab Treated Patients
Acronym: iCAMMS-IST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Anthony Traboulsee, Principal Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H10-02482; 142402 (Other: Health Canada - NOL)
Record Dates: First submitted 2011-01-26; First posted 2011-03-02 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; Relapsing Remitting Multiple Sclerosis; RRMS; Alemtuzumab; Demyelination; Remyelination; Tolerogenic; T cells; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Demyelinating Diseases; Autoimmune Diseases; Immune System Diseases
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Demyelinating Diseases; Demyelinating Autoimmune Diseases, CNS; Autoimmune Diseases of the Nervous System; Nervous System Diseases; Autoimmune Diseases; Immune System Diseases | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MabCampath-1h (Experimental): Single arm, single cohort study, all subjects will be dosed with alemtuzumab.
  Interventions: Drug: MabCampath-1h

INTERVENTIONS:
Drug: MabCampath-1h — Drug:10 mg/mL alemtuzumab intravenous infusion. Form: Sterile, clear, colorless solution. Dosage: 2 cycles. Month 0 dosed over 5 consecutive days; month 12 dosed over 3 consecutive days.
  Other Names: Alemtuzumab

SUMMARY:
There are two parts to this investigator sponsored trial (IST):

1. To perform advanced serial MRI studies on patients initiating alemtuzumab therapy.
2. To provide serum samples for the University of Southern California (USC) ICAM125 lymphocyte recovery study.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is an inflammatory demyelinating disease of the Central Nervous System (CNS). There are many forms of MS; although the majority are Relapsing Remitting (RRMS) representing approximately 80% of the cases. The disease appears to be more inflammatory in RRMS as manifested by an increase in Gadolinium (Gd) enhancement on MRI and an increase in inflammatory bio-assay markers.

Alemtuzumab; a humanized monoclonal antibody that targets the CD52 molecule present on T and B lymphocytes, natural killer (NK) cells, and monocytes and macrophages; effects rapid and sustained lymphocyte depletion and is approved for the treatment of B-cell chronic lymphocytic leukemia in many countries under the names CAMPATH or MabCAMPATH.

There are two parts to this Investigator Sponsored Trial (IST):

1. To perform advanced serial MRI studies on patients initiating alemtuzumab therapy.
2. To provide serum samples for the University of Southern California (USC) ICAM125 lymphocyte recovery study.

ELIGIBILITY:
Inclusion Criteria:

* Signed, informed consent form
* Age 18 to 50 years old (inclusive)
* Diagnosis of MS per update of McDonald criteria, and cranial MRI scan demonstrating white matter lesions attributable to MS within 10 years of screening
* Onset of MS symptoms within 15 years of screening
* Neurostatus (EDSS) score 0.0 to 5.0 (inclusive)
* 2 MS attacks (first episode or relapse) occurring in the 24 months prior to screening, with 1 attack in the 12 months prior to screening, with objective neurological signs confirmed by a physician.

Exclusion Criteria:

* Received prior therapy for MS other than corticosteroids within 28 days of screening; e.g., interferon's, IV immunoglobulin, and glatiramer acetate
* Exposure to natalizumab within 6 months of screening
* Any prior exposure to mitoxantrone, mycophenolate mofetil, azathioprine, cladribine, cyclophosphamide, cyclosporine A, methotrexate, rituximab, or any other immunosuppressive agent other than systemic corticosteroid treatment
* Has any progressive form of MS
* History of malignancy (exception for basal cell skin carcinoma)
* Previous hypersensitivity reaction to other immunoglobulin product
* Intolerance of pulsed corticosteroids, especially a history of steroid psychosis
* CD4+, CD8+, or CD19+ (i.e., absolute CD3+CD4+, CD3+CD8+, or CD19+/mm3) count <LLN at Screening; if abnormal cell count(s) return to within normal limits, eligibility may be reassessed
* Seropositivity for human immunodeficiency virus (HIV)
* Significant autoimmune disease (e.g, immune cytopenias, rheumatoid arthritis, systemic lupus erythematosus, other connective tissue disorders; vasculitis; inflammatory bowel disease; severe psoriasis)
* Presence of anti-thyroid stimulating hormone (TSH) receptor (TSHR) antibodies
* Active infection
* Latent tuberculosis unless effective anti-tuberculosis therapy has been completed, or active tuberculosis.
* Infection with hepatitis B virus or hepatitis C virus
* Of childbearing potential with a positive serum pregnancy test
* Unwilling to agree to use a reliable and acceptable contraceptive method throughout the study period
* Major psychiatric disorder that is not adequately controlled by treatment
* Epileptic seizures that are not adequately controlled by treatment
* Major systemic disease or other illness that would, in the opinion of the Investigator, compromise patient safety or interfere with the interpretation of study results
* Medical, psychiatric, cognitive, or other conditions
* Confirmed platelet count the lower limit of normal (LLN) of the evaluating laboratory at Screening or documented at 100,000/L within the past year on a sample without clumping
* Prior history of invasive fungal infections
* Cervical high risk human papilloma virus (HPV) positivity or abnormal cervical cytology other than abnormal squamous cells of undetermined significance (ASCUS).
* Seropositive for Trypanosoma cruzi or the Human T-lymphotropic virus type I or type II (HTLV-I/II) (testing required in endemic regions only)
* Any other illness or infection (latent or active) that, in the Investigator's opinion, could be exacerbated by alemtuzumab treatment
* Any hepatic or renal function value grade 2 or higher at Screening, with the exception of hyperbilirubinemia due to Gilbert's syndrome.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2011-03; Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Changes in normal appearing white matter from baseline through month 24. | 24 months
  The MRI study is designed to identify possible mechanisms by which alemtuzumab acts to protect the brain from inflammation and how it may enhance repair through remyelination.

SECONDARY OUTCOMES:
To identify specific changes in T cell subsets and functions in Relapsing Remitting Multiple Sclerosis from baseline through month 48. | 48 months
  Analyzing changes is immune responsiveness may reveal critical information about the mechanisms by which alemtuzumab acts, confirm the importance of specific immune cell types or molecules as targets for alemtuzumab treatment or may also be useful for monitoring drug effectiveness and safety.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Traboulsee, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] CAMMS223 Trial Investigators; Coles AJ, Compston DA, Selmaj KW, Lake SL, Moran S, Margolin DH, Norris K, Tandon PK. Alemtuzumab vs. interferon beta-1a in early multiple sclerosis. N Engl J Med. 2008 Oct 23;359(17):1786-801. doi: 10.1056/NEJMoa0802670. PMID 18946064
- [Background] Coles AJ, Cox A, Le Page E, Jones J, Trip SA, Deans J, Seaman S, Miller DH, Hale G, Waldmann H, Compston DA. The window of therapeutic opportunity in multiple sclerosis: evidence from monoclonal antibody therapy. J Neurol. 2006 Jan;253(1):98-108. doi: 10.1007/s00415-005-0934-5. Epub 2005 Jul 27. PMID 16044212
- [Derived] Gilmore W, Lund BT, Li P, Levy AM, Kelland EE, Akbari O, Groshen S, Cen SY, Pelletier D, Weiner LP, Javed A, Dunn JE, Traboulsee AL. Repopulation of T, B, and NK cells following alemtuzumab treatment in relapsing-remitting multiple sclerosis. J Neuroinflammation. 2020 Jun 15;17(1):189. doi: 10.1186/s12974-020-01847-9. PMID 32539719